CLINICAL TRIAL: NCT07294521
Title: Efficacy of Platelet-rich-Fibrin Gel in Patients With Chronic Leg Ulcers
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ahsan Tameez-ud-din, Registrar Dermatology, Pak Emirates Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERM112025
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Chronic Leg Ulcer
Keywords: Chronic leg ulcer; Platelet rich fibrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRF group (Experimental): Enrolled patients with chronic leg ulcers who will be administered PRF gel
  Interventions: Biological: Platelet rich Fibrin (PRF)

INTERVENTIONS:
Biological: Platelet rich Fibrin (PRF) — PRF is derived solely from the patient's own blood and does not contain any non-autologous additives, such as anticoagulants or bovine thrombin, as first-generation platelet concentrates (like some forms of PRP)

SUMMARY:
Platelet rich Fibrin (PRF) gel is an emerging as a novel treatment option for chronic leg ulcers and has the potential to become the 1st line option in these conditions. The objective of our study will be to assess the efficacy of PRF gel dressing in patients with non-infective chronic leg ulcers.

DETAILED DESCRIPTION:
Chronic leg ulcers (CLU) affect approximately 1% of the adult population and the prevalence increases significantly with age. The causes of CLU are mainly non-infective and include neuropathy, venous and arterial disease followed by less common causes like metabolic and hematological disorders. Leg ulcers severely impact the patients' quality of lives and frequently result in impaired mobility and financial dependence. There are several validated tools for the objective assessment of the ulcer severity. Bates Jensen wound assessment tool (BWAT) is one of these measures which will be originally developed for assessing pressure wounds but has been validated for other wounds such as CLU. BWAT consists of 13 scored items and can be used as a comprehensive tool for initial assessment as well as an indicator of treatment response.

The management is mainly supportive and depends on the underlying aetiology but there is a dearth of targeted wound management options that promote healing. Platelet rich Fibrin (PRF) gel is an emerging as a novel treatment option for chronic leg ulcers and has the potential to become the 1st line option in these conditions . The objective of our study will be to assess the efficacy of PRF gel dressing in patients with non-infective chronic leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* All male and female patients more than 35 years old with Chronic Leg Ulcers, presenting to the OPD will be included.

Exclusion Criteria:

* Patients with clinical signs of infected ulcers, patients in sepsis and immunosuppressed individuals will be excluded.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
50% improvement in Bates Jensen wound assessment tool (BWAT) score | 1 months
  Bates Jensen wound assessment tool (BWAT) is one of these measures which will be originally developed for assessing pressure wounds but has been validated for other wounds such as Chronic leg Ulcer. BWAT consists of 13 scored items and can be used as a comprehensive tool for initial assessment as well as an indicator of treatment response. The score ranges from 9 to 65 with higher scores mean worse healing (tissue degeneration), lower scores indicate improvement (regeneration).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Moizza Tahir, MBBS, FCPS, FRCP, Principal Investigator — Pak Emirates Military Hospital
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers as a general rule but during the publication process, it may be shared on editorial demand/ reviewer's comments in order to prove the authenticity of the data.